CLINICAL TRIAL: NCT05144438
Title: Prospective Evaluation of the Effectiveness of a Counseling Protocol to Reduce the Level of Exposure to Metallic Trace Elements (ETM)
Brief Title: Advice Protocol to Reduce the Level of Exposure to Metallic Trace Elements (ETM)
Acronym: ETM
Status: Completed | Type: Observational
Sponsor: Elsan (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01954-35
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Metallic Trace Elements; Metal-type Environmental Pollutants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women or woman in desire for conception: Towseek test : hair taking different questionnaires : environmental questionnaire, compliance questionnaire
  Interventions: Diagnostic Test: Toxseek test

INTERVENTIONS:
Diagnostic Test: Toxseek test — Hair taking

SUMMARY:
A French company (Toxseek, France, has developed a scientifically validated screening test based on a capillary determination of pollutants on a 3 cm lock of hair. The results of this screening allow physicians to discuss with their patients the question of environmental health and provide them with personalized behavioral advice in an attempt to eliminate the source of the pollutants identified.The main objective of the study is to assess the effectiveness of behavioral counseling on reducing the level of exposure to metal-type environmental pollutants (MTE) in pregnant women or women planning to have children.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Patient with desire to conceive
* 1st trimester of pregnancy
* Patient having been informed of the study and not opposing the use of the data collected
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Women under 18 years old
* 2nd and 3rd trimester of pregnancy
* Patient objecting to the use of the data collected
* Protected patient: adult under tutorship, curatorship or other protection legal, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women, over 18 years old, pregnant (first trimester) or desires conception
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who reduced their level of exposure within 4 months of metal avoidance advice. | 4 months
  The patient will be considered "successful" for the reduction of the exposure level, if all the metals with a "risky" exposure level during the 1st screening have gone to an exposure level "to be monitored" or "acceptable" during the 2nd screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle médical Saint Bernard, Saint-Rémy-de-Provence, France